CLINICAL TRIAL: NCT01509560
Title: PhaseII,Open-label,Pilot Study Evaluating the Safety+Efficacy of Certican ® in the Prevention of Chronic Graft-versus-host Disease+Late Pulmonary Complications After Allogeneic Hematopoietic Cell Transplantation Blood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Collaborators: Deutsche Klinik fuer Diagnostik (Other); ClinAssess GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ev02 (Everolimus-GvHD); 2010-023630-24 (EudraCT Number)
Record Dates: First submitted 2012-01-03; First posted 2012-01-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Condition After Allogenic Peripheral Stem Cell Transplantation (SCT)
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental): All patients will be given everolimus and the magnitude of the side effects will be measured
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Start therapy: 2x 0.75 mg/day (morning and evening) to receive a serum trough level of 3 - 5 ng/ml. First evaluation of Everolimus serum level 3-7 days after start of therapy, second 7 days later, subsequently on study weeks 4, 6, 9, 12 and 16. Dose has to be adapted if trough level exceeds 5 ng/ml. As soon as Everolimus trough level exceeds 3 ng/ml after start of therapy, calineurine inhibitors (e.g. cyclosporine) will be reduced: halve of the dose for the 3 consecutive days, withdrawal on day 4.
  Prednisone will be reduced accordingly (a 22 weeks scheme is recommended) Everolimus will be used for 98 days or 14 weeks, as described above Everolimus therapy might be extended (independently of the study) if the patient suffering from milde chronic GvHD (according to NIH criteria) or milde PTOLD and lung function score is not reduced more than 25% since begin of Everolimus therapy Everolimus will be reduced to 50% of the dosage for 2 weeks before withdraw (normally weeks 15 and 16
  Other Names: Everolimus: Certican®

SUMMARY:
In this prospective study is to examine whether the use of everolimus in patients after allogeneic SCT as part of GVHD prophylaxis for a further review in clinical studies is appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients after allogeneic stem cell transplantation aged ≥ 18 years
* Prophylaxes of GvHD with calcineurin inhibitors (Ciclosporine A, Tacrolimus) and MTX or MMF (previous therapy of acute GvHD with additional prednisone is permitted)
* Increased risk of chronic GvHD, defined by
* Male with female donor
* HLA mismatch class I- or II towards GvHD
* Persistant active acute GvHD on day +50 after stem cell transplantation despite of high-dose steroids and cyclosporine
* Reduction of baseline FEV1 or DLCO (examined 0 - 50 days before transplantation) of ≥ 25%
* New occurrence of acute GvHD between day +50 and +100 after stem cell transplantation
* Informed concent

Exclusion Criteria:

* Use (prophylactic or therapeutic) of mTor inhibitors after SCT
* Overlap of acute and chronic GvHD
* Total cholesterol ≥ 3-fold of upper limit (UL) or triglycerides ≥ 3-fold UL
* GOT, GPT, Bilirubin ≥ 3-fold UL (if not related to GvHD)
* Creatinine ≥ 3-fold UL
* Confirmed active hepatitis B or C
* All circumstances where impaired wound healing might be a risk factor, esp. surgical interventions in the last weeks, ulcers of skin or mucosa
* Known intolerance to Everolimus, Sirolimus or other compoments of Certican®
* Lactose intolerance
* Pregnancy or lactation
* Women in reproductive age, except of women with the following criteria:
* Postmenopausal (12 month natural amenorrhea)
* Postoperativ (≥ 6 months after bilateral ovariectomy with / without hysterectomy)
* During therapy and at least 6 months after the last application of Everolimus: regular and correct high-effective contraception (Pearl-Index < 1; e. g. oral contraception, intrauterine device, implantate, contraceptive patch, combination of barrier methods (condom and cervical cap/diaphragm), abstinence
* Men, not using one of the following methods of contraception during therapy and at least 6 month after the last application of Everolimus:
* Sexual abstinence
* Vasectomy
* Condom
* Impairments or diseases reducing the ability of informed consent
* Participation of another study (e.g. for prophylactic immunsuppression in the stem cell transplantation procedure) within the last 60 day before recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Frequency of early withdrawal of treatment within the first 6 weeks on Everolimus | 16 months
  Primary endpoint Frequency of early withdrawal of treatment within the first 6 weeks on Everolimus
  Reasons for withdrawal of Everolimus treatment:
  * Unacceptabel toxicity
  * Therapy failure:
  * Recurrence of moderate or severe chronic GvHD (according to NIH criteria), clearly differentiated from acute forms of GvHD
  * Reduction of LFS of more than 25% compared to the last value within 14 days before Everolimus treatment
  * Therapy with immunosuppressive drugs in addition to Everolimus

SECONDARY OUTCOMES:
Adverse drug reactions on Everolimus | 16 months
  * Adverse drug reactions on Everolimus
  * Frequency and grading of GvHD (according to NIH concerns) and POLT
  * Lung function score (LFS)
  * Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schleuning, Prof. Dr. med., Principal Investigator — Stiftung Deutsche Klinik für Diagnostik GmbH
Locations (1):
- Zentrum für Knochenmark- und Blutstammzelltransplantation,, Wiesbaden, Hesse, Germany